CLINICAL TRIAL: NCT04731402
Title: The Effect of Acupressure, Laughter Yoga and Conscious Awareness on Menopausal Symptoms and Quality of Life in Menopausal Women.
Brief Title: The Effect of Acupressure, Laughter Yoga and Mindfulness on Menopausal Symptoms and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hacer Unver, PhD, phd, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: inonu university ethics
Record Dates: First submitted 2021-01-12; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Menopausal Symptoms; Quality of Life
MeSH Terms: interventions — Acupressure; Laughter Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acupressure (Experimental): Acupressure group Acupressure application will be applied twice a week, 24 times in total in 12 weeks. Each acupressure point will be massaged for 30 seconds to provide circulation before compression. After the massage, pressures will be applied consecutively for 90 seconds. The session duration for each woman will be 8 minutes in total, with 2 minutes for each point in each attempt.
  Interventions: Other: Acupressure, laughter yoga and mindfulness stress reduction program
- Laughter Yoga (Experimental): Laughter Yoga group Laughter yoga sessions begin with gentle warm-up techniques that include stretching and stretching movements, songs, applause, and body movements. Therapy sessions are between 30-45 minutes.8 sessions of laughter yoga will be done once a week.
  Interventions: Other: Acupressure, laughter yoga and mindfulness stress reduction program
- mindfulness stress reduction program (Experimental): mindfulness stress reduction program mindfulness stress reduction program consists of 8 weeks. each week is 2.5 hours. each week has a different theme. There is a 6-hour silence day in the 6th week of the program.
  Interventions: Other: Acupressure, laughter yoga and mindfulness stress reduction program
- Control Group (No Intervention): INTERVENTION NOT IMPLEMENTED

INTERVENTIONS:
Other: Acupressure, laughter yoga and mindfulness stress reduction program — Initiatives will be applied to the experimental group. only measurement tools will be applied to the control group
  Arms: Acupressure; Laughter Yoga; mindfulness stress reduction program

SUMMARY:
The aim of the study is to determine the effect of acupressure, laughter yoga and Mindfulness stress reduction program on menopausal symptoms and quality of life.Menopausal period, which is one of the life stages, causes physiological changes and can decrease the quality of life.

The research is a randomized controlled trial. 180 women who meet the conditions for research will be included in the study. Three instruments were used to obtain the research data: Personal Information Form,Menopausal Symptoms Rating Scale and Menopause-Specific Quality of Life Scale.

DETAILED DESCRIPTION:
On average, one third of a woman's life passes during menopause. The menopausal period is an important period that brings many physical and psychological changes with it and significantly affects the disease process and the family and society. Cultural and ethnic characteristics of the society are among the important factors that affect women's attitudes towards menopause and the meaning of middle age for women.women seek ways to deal with menopausal symptoms.

women prefer drug-free coping methods. Mindfulness stress reduction program, yoga and laughter yoga are an alternative way to reduce menopausal symptoms.. These methods can reduce the complaints and increase the quality of life. For this reason, the effect should be determined in the menopausal period.

ELIGIBILITY:
Inclusion Criteria:

* in the menopausal period

Exclusion Criteria:

* presence of psychiatric illness using psychiatric medication

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It is a specific study for menopause
Enrollment: 180 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Acupressure, Laughter Yoga and mindfulness stress reduction program Effects on menopause symptoms | Up to 12 weeks
  Menopause Rating Scale is an 11 item scale.The five-point Likert type scale has three sub-dimensions.The higher the scores of each item, the higher the complaints, the higher the total score of the scale, the higher the menopausal complaints.
Acupressure, Laughter Yoga and mindfulness stress reduction program Effects on menopausal quality of life | Up to 12 weeks
  Menopausal Quality of Life Scale is a Likert-type scale with 29 questions and consists of four domains: vasomotor, psychosocial, physical and sexual. Each question score is from 0 to 6. The increase in the scale score indicates that the severity of the complaints increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacer, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No